CLINICAL TRIAL: NCT04743492
Title: How Pain Resilience Determines the Efficacy of Holistic Health Care of Patients With Migraine
Brief Title: Pain Resilience and Holistic Health Care of Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Changhua Christian Hospital (Other)
Collaborators: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y_109_0314
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-09

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CBT group (Experimental): cognitive behavioral therapy (CBT)+routine medical care
  Interventions: Behavioral: cognitive behavioral therapy
- exercise therapy group (Experimental): physiotherapy-exercise therapy+routine medical care
  Interventions: Behavioral: cognitive behavioral therapy
- breathe training group (Experimental): using biofeedback devices to train breathing speed+routine medical care
  Interventions: Behavioral: cognitive behavioral therapy
- usual care (No Intervention): accepting only routine medical care

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — cognitive behavioral therapy delivered by clinical psychologists in order to help patients gain coping skills.
  Arms: CBT group; breathe training group; exercise therapy group

SUMMARY:
The purpose of this study is to investigate how pain resilience (as a personality characteristic or a strength) moderate the efficacy of treatment for patients with migraine.

The primary objective of the current study is to explore the moderation effect of pain resilience between initial pain and the treatment outcome of the holistic healthcare programs. The investigators hypothesize that participants with higher level of pain resilience will show more improvements in the quality of life, less disability (assessed with the Migraine Disability Assessment Test, MIDAS), less frequency and lower severity of pain, and higher heart-rate variability after training. A secondary finding that can be obtained through the study is the comparison between the enhancement of heart rate variability in participants receiving different kinds of non-pharmacological therapies.

DETAILED DESCRIPTION:
Introduction：A multi-national research that included data from Taiwan found that chronic headache is one of the top two disorders (alongside with chronic low back pain) with the most patients having longest years of living with disabilities through year 1999 to 2017. It does not only impact a sufferer's ability to work, but also limit one's participation in a variety of daily housework, leisure activities, etc. Quality of life is also impacted. According to a systematic review on behavioral interventions for migraine, cognitive behavioral therapy (CBT) is one of the most common non-pharmacological practices implemented and studied. CBT has been found to be effective in reducing the intensity and frequency of headache, compared to waitlist controls. Another commonly discussed non-pharmacological treatment for migraine is exercise therapy.

In regard to the controversial findings from therapeutic clinical trials, the unsolved puzzle is: why do some show improvements while the others remained unchanged or worse? It is found that psychological resilience for pain can be a determining factor in task persistence despite the interruption of pain. Pain resilience specifically refers to the cognitive and behavioral aspects of an individual when one is trying to deal with pain. In a study investigating negative pain beliefs (i.e. fear avoidance and pain catastrophizing) and pain outcomes (functional and movement aspects), pain resilience was found to moderate the relationship between pain beliefs and pain outcomes. The authors found that only in individuals with low level of pain resilience was the negative pain beliefs related to greater movement-relate pain. Since pain resilience is such an important capacity/ dynamic process in coping with chronic pain, the current study aims at investigating how pain resilience can be a moderating factor determining the outcome of pain management in patients with migraine.

Objectives：The primary objective of the current study is to explore the moderation effect of pain resilience between initial pain and the treatment outcome of the holistic healthcare programs. The investigators hypothesize that participants with higher level of pain resilience will show more improvements in the quality of life, less disability (assessed with MIDAS), less frequency and lower severity of pain, and higher heart-rate variability after training. A secondary finding that can be obtained through the study is the comparison between the enhancement of heart rate variability in participants receiving different kinds of non-pharmacological therapies.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with migraine

Exclusion Criteria:

* uncontrolled hypertension
* coronary artery disease
* arrhythmia
* secondary headache(except for medication overuse headache)a
* age under 20

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
level of disability | 8 weeks
  Measured with the Migraine Disability Assessment Test (MIDAS). The total score ranges from 0 to 21 or more. Higher score indicates more disabilities related to migraine. Score over 21 indicates severe disability.
severity of pain | 8 weeks
  Self-reported pain scores range from 0 to 10, with 0 meaning no pain at all, and 10 meaning extreme pain. Scoring over 7 indicates severe pain.

SECONDARY OUTCOMES:
heart rate variability | 8 weeks
  measured with wearable devices

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Jun Liu, MSc, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Chang-hua, Taiwan

IPD SHARING:
Plan to Share IPD: No